CLINICAL TRIAL: NCT00771914
Title: The Effects of Omega-3 Fatty Acids on Aspirin Resistance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: GlaxoSmithKline (Industry); American College of Clinical Pharmacy (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Robert Block, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Study Protocol 112421
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Increased Drug Resistance
Keywords: aspirin; omega 3 fatty acids; Lovaza; myocardial infarction; aspirin resistance; cardiovascular disease
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases | interventions — Aspirin; Omacor; Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza (Experimental): First Placebo, then 4 grams of Lovaza, then 81mg of Aspirin, then both 4 grams of Lovaza and 81 mg of Aspirin
  Interventions: Drug: Aspirin; Drug: Lovaza; Drug: Both Aspirin and Lovaza; Other: Placebo
- Aspirin, Lovaza, Both Aspirin and Lovaza, Placebo (Experimental): First 81mg of Aspirin, then 4 grams of Lovaza, then both 81mg of Aspirin and 4 grams of Lovaza, then placebo
  Interventions: Drug: Aspirin; Drug: Lovaza; Drug: Both Aspirin and Lovaza; Other: Placebo
- Lovaza, Both Aspirin and Lovaza, Placebo, Aspirin (Experimental): First 4 grams of Lovaza, then both 81mg of Aspirin and 4 grams of Lovaza, then placebo, then 81mg of Aspirin
  Interventions: Drug: Aspirin; Drug: Lovaza; Drug: Both Aspirin and Lovaza; Other: Placebo
- Both Aspirin and Lovaza, Placebo, Lovaza, Aspirin (Experimental): First both 81mg of Aspirin and 4 grams of Lovaza, then placebo, then 4 grams of Lovaza, then 81mg of Aspirin
  Interventions: Drug: Aspirin; Drug: Lovaza; Drug: Both Aspirin and Lovaza; Other: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin 81mg tablet
Drug: Lovaza — Lovaza 4 grams
  Other Names: ethyl EPA + DHA; fish oil
Drug: Both Aspirin and Lovaza — Lovaza 4 grams plus aspirin 81 mg
  Other Names: Lovaza and aspirin
Other: Placebo — Capsule resembling fish oil and a tablet resembling aspirin

SUMMARY:
The purpose of this study is to determine if omega-3 fatty acids enhance the antiplatelet effects of aspirin.

DETAILED DESCRIPTION:
Although aspirin has been a stalwart treatment in the prevention and treatment of myocardial infarction and stroke, it does not have its expected effects in a significant proportion of the population. This phenomenon has been termed "aspirin resistance". Omega-3 fatty acid supplementation has been associated with a reduced risk of sudden cardiac death and myocardial infarction. The beneficial effects of omega-3s are considered to be partially due to their ability to prevent platelet aggregation. However, the ability of omega-3s to enhance the effects of aspirin in those who suffer from aspirin resistance has not been determined. It is known that aspirin stimulates the production of potent lipid mediators from omega-3 fatty acids and that these mediators have powerful antiinflammatory and tissue-protective effects. Thus, the treatment of individuals at high risk for myocardial infarction and stroke with both aspirin and a pharmaceutical-grade omega-3 fatty acid medication may be a powerful combination in the prevention and treatment of life-threatening cardiovascular disease.

Study Protocol: Non-smoking male and female subjects between the ages of 18 and 50 not taking any medications, vitamin pills, nutritional supplements, or herbal preparations were recruited. Subjects with a history of chronic diseases (e.g. cardiovascular, renal, hepatic, neurodegenerative, neoplastic, metabolic {diabetes}, hypertension; based on screening medical history, a complete blood count, and comprehensive metabolic profile), or allergic reactions to aspirin, fish, fish oils, or non-steroidal anti-inflammatory drugs were excluded. Other exclusions included drinking more than three alcoholic beverages a day, or having any of the following conditions: an ulcer or bleeding in the stomach, liver or kidney disease, bleeding or blood clotting disorder (e.g. hemophilia), congestive heart failure, fluid retention, high blood pressure, gout, asthma, arthritis, or nasal polyps. This was a randomized, placebo-controlled, double-blinded trial with a cross-over design. Each subject served as his/her own control. The study involved four visits four weeks apart, all hosted in the University of Rochester Clinical Research Center. At each separate study visit, each subject received (using a randomized protocol) placebo, 81 mg aspirin, 4 g Lovaza(R)(3.4g of EPA+DHA), or both aspirin and Lovaza(R). Thus, each subject received each of these treatments individually in a random fashion over the four visits. Subjects, Center staff, and investigators were blinded as to which treatment was given at each visit and this ensured by the study pharmacist making the tablets and capsules for each treatment appear identical. Prior to each visit, subjects ate a standard low-fat dinner the prior evening, then fasted for at least 8 hours prior to arrival at the Center. Subjects were required to abstain from taking aspirin or non-steroidal anti-inflammatory drugs for 10 days prior to each visit and omega-3 fatty acids for 30 days prior to the baseline study visit, and all subsequent clinic visits. Visits lasted approximately 6 hours, with subjects at bedrest. A venous catheter was placed in a peripheral vein (saline lock, 18 gauge or larger, {no heparin used} in the forearm) with blood drawn, at baseline and 4 hours post-treatment, into citrated tubes at each visit for Platelet Function Analyzer-100 (PFA-100-Siemens, Deerfield, IL) closure time testing. Subjects were provided with a standard low-fat breakfast after the baseline phlebotomy.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate by providing informed consent and committing to complete the study. This includes adhering to the study diet.
* No chronic disease by history and based on a complete blood count and comprehensive metabolic profile.
* Commitment to not taking aspirin, non-steroidal anti-inflammatory medications, and to limit fish intake to ≤2 meals during the 7 days prior to each CRC study period. They will also need to abstain from taking a list of over-the-counter medications that include aspirin. For the duration of the study, they will also be asked to abstain from taking fish and flax seed oil supplements.

Exclusion Criteria:

* Reports the presence of chronic disease (e.g. cardiovascular, renal, hepatic, neurodegenerative, neoplastic, metabolic {diabetes}, hypertension).
* Reports taking a systemic medication chronically.
* History of serious adverse reaction or allergy to aspirin or fish oil.
* Baseline platelet count <100 000 or >500 000, hematocrit <30%, or white blood cell count >20 000.
* Any abnormality from a screening CBC and complete blood count that suggests acute or chronic disease.
* Nicotine user.
* History of alcohol abuse
* Pregnancy by history or urine/serum pregnancy test
* History of intestinal malabsorption syndrome including gastric bypass surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Block, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester School of Medicine and Dentistry, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza: First Placebo, then 4 grams of Lovaza, then 81mg of Aspirin, then both 81mg of Aspirin and 4 grams of Lovaza
- Aspirin, Lovaza, Both Aspirin and Lovaza, Placebo: First 81mg of Aspirin, then both 81mg of Aspirin and 4 grams of Lovaza, then 4 grams of Lovaza, then 81mg of Aspirin
- Lovaza, Both Aspirin and Lovaza, Placebo, Aspirin: First 4 grams of Lovaza, then both 81mg of Aspirin and 4 grams of Lovaza, then placebo, then 81 mg of Aspirin
Period: Overall Study
Arm/Group | Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza | Aspirin, Lovaza, Both Aspirin and Lovaza, Placebo | Lovaza, Both Aspirin and Lovaza, Placebo, Aspirin | Both Aspirin and Lovaza, Placebo, Lovaza, Aspirin
Started | 7 | 6 | 6 | 8
Completed | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza: First Placebo, then 4 grams of Lovaza, then 81 mg of aspirin, then both 81mg of Aspirin and 4 grams of Lovaza
- Total: Total of all reporting groups
Arm/Group | Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza | Aspirin, Lovaza, Both Aspirin and Lovaza, Placebo | Lovaza, Both Aspirin and Lovaza, Placebo, Aspirin | Both Aspirin and Lovaza, Placebo, Lovaza, Aspirin | Total
Number analyzed (Participants) | 7 | 6 | 6 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 6 | 8 | 27
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.7 (9.7) | 32.9 (11.6) | 25.9 (3.4) | 29.3 (10.2) | 29.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 4 | 14
  Male | 3 | 3 | 3 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 6 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: the Difference Between the Time to Clot Formation in Seconds at Baseline and After Each Treatment
Description: The PFA-100 test measures platelet function as the time that it takes for a clot to form in a collagen-lined cartridge.
Time Frame: 4 hours
Population: Each participant acted as own control since each received the intervention (placebo, aspirin, lovaza, and both aspirin and lovaza) and had these effects compared to baseline (four hour effect of each intervention).
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Placebo: All participants received Placebo intervention regardless of sequence.
- Aspirin: All participants received Aspirin intervention regardless of sequence.
- Lovaza: All participants received Lovaza intervention regardless of sequence.
- Both Aspirin and Lovaza: All participants received Aspirin and Lovaza intervention regardless of sequence.
Arm/Group | Placebo | Aspirin | Lovaza | Both Aspirin and Lovaza
Number analyzed (Participants) | 25 | 25 | 25 | 25
seconds | 0.0 (30) | 10.9 (50.23) | -6.5 (63.6) | 30.5 (60.3)
Statistical Analysis 1: Comparison: Placebo; The Wilcoxon Signed-Rank Test was used to determine significant differences between the closure time effect (clotting)in seconds from baseline compared to four hours after placebo; Test type: Superiority or Other; p = 0.00, Wilcoxon (Mann-Whitney) — The analyses were not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.00
Statistical Analysis 2: Comparison: Placebo vs Aspirin; The Wilcoxon Signed-Rank Test was used to determine significant differences between the closure time effect (clotting)in seconds from Aspirin compared to Placebo; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney) — The analyses were not adjusted for multiple comparisons; Median Difference (Final Values) = 12
Statistical Analysis 3: Comparison: Placebo vs Lovaza; The Wilcoxon Signed-Rank Test was used to determine significant differences between the closure time effect (clotting)in seconds from Lovaza compared to Placebo; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney) — The analyses were not adjusted for multiple comparisons; Mean Difference (Final Values) = -8
Statistical Analysis 4: Comparison: Placebo vs Both Aspirin and Lovaza; The Wilcoxon Signed-Rank Test was used to determine significant differences between the closure time effect (clotting)in seconds from both Aspirin and Lovaza compared to Placebo; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney) — The analyses were not adjusted for multiple comparisons; Mean Difference (Final Values) = 30

ADVERSE EVENTS:
Arm/Group | Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza | Aspirin, Lovaza, Both Aspirin and Lovaza, Placebo | Lovaza, Both Aspirin and Lovaza, Placebo, Aspirin | Both Aspirin and Lovaza, Placebo, Lovaza, Aspirin
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3.85% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Lovaza, Aspirin, Both Aspirin and Lovaza (N=7) | Aspirin, Lovaza, Both Aspirin and Lovaza, Placebo (N=6) | Lovaza, Both Aspirin and Lovaza, Placebo, Aspirin (N=6) | Both Aspirin and Lovaza, Placebo, Lovaza, Aspirin (N=6)
Headache, nausea, lightheadness (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No